CLINICAL TRIAL: NCT05174676
Title: Robotic Enhanced Error Training of Upper Limb Function in Post-stroke Patients: A Randomized Controlled Trial
Brief Title: Robotic Enhanced Error Training of Upper Limb Function in Post-stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reuth Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0012-21-RRH
Record Dates: First submitted 2021-11-29; First posted 2022-01-03 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: CVA (Cerebrovascular Accident); Paresis
Keywords: Brain plasticity; Upper limb function; Robotic rehabilitation; Error augmentation or enhancement
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The participant will receive 6 therapy sessions of approximately 25 minutes each WITH the application of error enhancement.
  Interventions: Device: Dextreme
- Control (Sham Comparator): The participant will receive 6 therapy sessions of approximately 25 minutes each WITHOUT the application of error enhancement.
  Interventions: Device: Dextreme

INTERVENTIONS:
Device: Dextreme — A unique robotic device capable of applying motor error enhancement forces during upper limb practice in a virtual environment. The forces stimulate the body's instinctive adaptive response, which does not require the use of cognition to correct the movement.
  The setting of stroke patients in a simulated environment enhances patient motivation and participation. The completion of "games" (tasks) is a great indicator for the patients that they are progressing in the treatment and are on their way to recovery.

SUMMARY:
Background: Stroke is a common cause of morbidity, including paresis, and stroke survivors often have reduced function in their paretic arm. Many do not regain full recovery of their arm function, which negatively impacts their quality of life. Recent studies have indicated that robotic training may improve upper limb function abilities among stroke survivors, by enabling repetitive, adaptive, and intensive training and more accurate control of task complexity. Robotic training in addition to standard rehabilitative care has shown promise for improving functional skills among stroke survivors. One type of robotic training is error enhancement, whereby an error made by the patient is exaggerated, increasing the signal to noise ratio which causes errors to be more noticeable. This, in turn, enhances movement correction. Previous studies have found that error enhancement has promise as a clinical treatment for patients with motor deficits.

Objectives: This study aims to evaluate the effect of a robotic device (DeXtreme) on the functional capabilities of the paretic arm of stroke survivors. This device aims to improve arm function by utilizing error enhancement techniques.

Methods: A double-blind randomized placebo-controlled study comparing treatment outcomes between two groups to assess the effect of error enhancement robotic training on functional use of the arm and hand in patients after stroke. Forty stroke patients will undergo 6 sessions of 25 minutes each with the Dextreme device. One group will receive training with error enhancement forces applied, while the control group will receive similar training without error enhancement. Outcomes (motor function, speed, tone, and spasticity) will be assessed twice prior to and following the treatment sessions,

DETAILED DESCRIPTION:
Background: At least 85% of stroke survivors suffer from weakness in their upper limbs. Around 40% of stroke survivors will suffer from severe handicap in their paretic arm, negatively affecting their independence and quality of life. Only 30% - 70% of survivors will recover enough function to enable daily use of the arm. These numbers clearly indicate that despite significant advances in the ability to rehabilitate stroke patients, there is still a need for more effective methods.

Traditional rehabilitative methods to improve arm function after stroke are often time-consuming and labor-intensive. Only few of these methods induce slightly improved arm function, and full recovery of arm function is often not achieved. Recently, studies have indicated that robotic training has promise for improving functional abilities among stroke survivors, by enabling repetitive, adaptive, and intensive training and more accurate control of task complexity. One type of robotic training that is particularly promising is error enhancement, which utilizes the adaptive capabilities of the nervous system to improve motor function.

Study Objectives: To examine the change in the upper limb function among stroke patients undergoing error enhancement treatment compared to a control group in the following domains:

1. Motor Function (Motor Assessment Scale-MAS, Fugl-Meyer Assessment)
2. Speed (Box and Blocks Assessment)
3. Tone and Spasticity (Modified Ashworth Scale)

Methods Participants: 40 stroke patients with hemiparesis recruited 21-60 days following the Cerebrovascular accident event.

Recruitment: Electronic medical records of newly hospitalized patients will be screened to identify potential study participants. Participation will be offered to each patient who meets the study inclusion criteria. After obtaining informed consent, an intake session will take place for both participant screening and evaluation, conducted by a qualified occupational therapist. Patients who successfully pass the intake screening session will undergo randomization to one of the two study arms.

Another occupational therapist will be conducting the treatment sessions. Patients in the intervention arm will undergo training sessions on the Dextreme robot device, while the error enhancement mechanism is switched on, while the patients in the control arm will undergo similar sessions with the mechanism switched off. A second patient assessment will be conducted within 96 hours following the last treatment session by an allocation-blinded occupational therapist.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew speaker.
* First stroke (ischemic or hemorrhagic).
* Weakness on one side of the body (left or right).
* At least 21 days have passed since the stroke event.
* At least 21 days left for inpatient rehabilitative care.
* Have partial mobility in the elbow and shoulder and the ability to open and close the hand.
* A minimum score of 10 (out of the 66) on the Fugl-Meyer Assessment for the upper limb.
* Cognitive status: Mini-Mental State Examination [MMSE] = 23 or higher; or MoCA test = 26 or higher.

Exclusion Criteria:

* Complete paralysis of the affected side.
* Comorbid central nervous system diseases that may affect brain plasticity (MS, ALS).
* Sensory Aphasia (as per the medical diagnosis).
* One-side neglect.
* Apraxia.
* Pregnancy or breastfeeding.
* Strong pain in the shoulder (VAS>6) that may prevent the ability to execute the tasks
* A severe orthopedic problem in the upper limb that prevents the ability to execute tasks on the robotic system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment #1 | 1 session up to 96 hours prior to first treatment session
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. This study will utilize the Fugl-Meyer Assessment only for the paretic upper limb. The assessment scores will range from 0 to 66, with a lower score indicating higher impairment. A minimum score of 10 will be set as an inclusion criterion.
Fugl-Meyer Assessment #2 | 1 session up to 96 hours after last (6th) treatment session
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. This study will utilize the Fugl-Meyer Assessment only for the paretic upper limb. The assessment scores will range from 0 to 66, with a lower score indicating higher impairment. A minimum score of 10 will be set as an inclusion criterion.
Motor Assessment Scale (MAS) #1 | 1 session up to 96 hours prior to first treatment session
  The Motor Assessment Scale (MAS) is a performance-based scale used to assess everyday motor function in patients with stroke. It is a validated tool comprised of 18 tasks for the upper limbs. Each task is given a score of 0 (unable to perform) to 1 (able to perform), and the overall score ranges from 0 to 18. This assessment will be applied to both upper limbs.
Motor Assessment Scale (MAS) #2 | 1 session up to 96 hours after last (6th) treatment session
  The Motor Assessment Scale (MAS) is a performance-based scale used to assess everyday motor function in patients with stroke. It is a validated tool comprised of 18 tasks for the upper limbs. Each task is given a score of 0 (unable to perform) to 1 (able to perform), and the overall score ranges from 0 to 18. This assessment will be applied to both upper limbs.
Box and Block Test (BBT) #1 | 1 session up to 96 hours prior to first treatment session
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including patients with stroke.
  During the assessment, the subject sits at a table in front of a box with two parts. The first part has 150 blocks, while the second part is empty. The participant must move as many blocks as he can (one at a time) in 60 seconds. The final score is the number of blocks he was able to move (out of a possible score of 150).
Box and Block Test (BBT) #2 | 1 session up to 96 hours after last (6th) treatment session
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including patients with stroke.
  During the assessment, the subject sits at a table in front of a box with two parts. The first part has 150 blocks, while the second part is empty. The participant must move as many blocks as he can (one at a time) in 60 seconds. The final score is the number of blocks he was able to move (out of a possible score of 150).
Modified Ashworth Scale #1 | 1 session up to 96 hours prior to first treatment session
  The Modified Ashworth Scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform. It is performed by extending the patient's limb from a position of maximal possible flexion to maximal possible extension. Afterwards, the patient is assessed while moving from extension to flexion.
Modified Ashworth Scale #2 | 1 session up to 96 hours after last (6th) treatment session
  The Modified Ashworth Scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform. It is performed by extending the patient's limb from a position of maximal possible flexion to maximal possible extension. Afterwards, the patient is assessed while moving from extension to flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Rami Mansour, MD, Principal Investigator — Reuth Rehabilitation Hospital
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No